CLINICAL TRIAL: NCT00027742
Title: A Phase II Study of Temozolomide (Temodar) and Peglated Interferon Alfa-2B (PEGIntron) in the Treatment of Advanced Melanoma
Brief Title: Temozolomide and Interferon Alfa in Treating Patients With Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 01-005; CDR0000069062 (Registry Identifier: PDQ (Physician Data Query)); NCI-G01-2031
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Intraocular Melanoma; Melanoma (Skin)
Keywords: iris melanoma; extraocular extension melanoma; recurrent intraocular melanoma; stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — Temozolomide

INTERVENTIONS:
Biological: pegylated interferon alfa
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Interferon alfa may interfere with the growth of cancer cells. Combining chemotherapy with interferon alfa may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining temozolomide and interferon alfa in treating patients who have stage III or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in patients with advanced melanoma treated with temozolomide and pegylated interferon alfa.
* Determine the toxicity profile of this regimen in these patients.
* Determine the duration of disease response and overall survival of patients treated with this regimen.

OUTLINE: Patients are stratified according to CNS metastases (yes vs no).

Patients receive oral temozolomide once daily on weeks 1-6 and pegylated interferon alfa subcutaneously once weekly on weeks 1-8. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 23-61 patients (12-35 without CNS metastases and 11-26 with CNS metastases) will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant melanoma

  * Unresectable stage III or stage IV disease
  * Ocular, mucosal, or cutaneous melanoma
* Measurable disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 150,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT/SGPT no greater than 3 times ULN
* Alkaline phosphatase no greater than 3 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No history of severe cardiovascular disease
* No myocardial infarction within the past 6 months
* No unstable angina
* No New York Heart Association class III or IV heart disease (congestive heart failure)
* No ventricular tachyarrhythmias

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No AIDS-related illness
* No frequent vomiting or other medical condition that would preclude oral medication intake (e.g., partial bowel obstruction)
* No serious infection requiring IV antibiotics
* No psychiatric disorder requiring ongoing therapy or medication
* No nonmalignant illness or other medical condition that would preclude study
* No other active malignancy within the past 2 years except non-melanoma skin cancer, carcinoma in situ of the cervix, or T1a or b prostate cancer detected initially during transurethral resection of the prostate (TURP) (comprising less than 5% of resected tissue) with PSA level normal since TURP

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior biologic therapy or immunotherapy and recovered
* No concurrent immunotherapy

Chemotherapy:

* No prior dacarbazine
* No prior temozolomide
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent systemic corticosteroids

Radiotherapy:

* At least 3 weeks since prior radiotherapy, interstitial brachytherapy, or radiosurgery
* At least 3 weeks since prior radiotherapy to the brain for brain metastases
* Prior radiotherapy to indicator lesions allowed if there is evidence of disease progression
* Recovered from prior radiotherapy
* No concurrent radiotherapy

Surgery:

* At least 2 weeks since prior surgical procedure requiring general anesthesia and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-05; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Jen Hwu, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Krown SE, Hwu WJ, Menell JH, et al.: A phase II study of temozolomide (TMZ) and pegylated interferon α-2b (PGI) in the treatment of advanced melanoma. [Abstract] J Clin Oncol 22 (Suppl 14): A-7533, 718s, 2004.